CLINICAL TRIAL: NCT04421456
Title: A Randomized, Double-blind, Parallel-group Trial to Investigate the Safety and Efficacy of GWP42003-P Versus Placebo as Adjunctive Therapy in Participants With Schizophrenia Experiencing Inadequate Response to Ongoing Antipsychotic Treatment
Brief Title: Trial to Investigate the Safety and Efficacy of GWP42003-P Versus Placebo as Adjunctive Therapy in Participants With Schizophrenia Experiencing Inadequate Response to Ongoing Antipsychotic Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated based on a business decision by the Sponsor.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWAP19030; 2019-003369-16 (EudraCT Number)
Record Dates: First submitted 2020-05-27; First posted 2020-06-09 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Schizophrenia
Keywords: GWP42003-P; adjunctive therapy; inadequate response to ongoing antipsychotic treatment
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GWP42003-P 300 mg (Experimental): GWP42003-P 300 milligrams (mg) per day
  Interventions: Drug: GWP42003-P
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo
- GWP42003-P 1000 mg (Experimental): GWP42003-P 1000 mg per day
  Interventions: Drug: GWP42003-P

INTERVENTIONS:
Drug: GWP42003-P — oral solution containing 100 milligrams per milliliter (mg/mL) cannabidiol (CBD) dissolved in the excipients sesame oil and anhydrous ethanol (10% v/v), with sweetener (sucralose), and strawberry flavoring
  Arms: GWP42003-P 1000 mg; GWP42003-P 300 mg
Drug: Placebo — oral solution containing the excipients sesame oil and anhydrous ethanol, with added β-carotene, sweetener (sucralose), and strawberry flavoring
  Arms: Placebo

SUMMARY:
This study will be conducted to evaluate the efficacy, safety, and tolerability of GWP42003-P versus placebo in participants with schizophrenia experiencing inadequate response to ongoing antipsychotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 55 years of age at the time of signing the Informed Consent Form (ICF)
* Willing and able to give informed consent for participation in the trial
* Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of schizophrenia, confirmed by the Mini International Neuropsychiatric Interview (MINI)
* Clinically stable outpatient
* Positive and Negative Symptoms Scale (PANSS) Total (PANSS-T) score of ≥ 60 and < 110 at screening and baseline visits
* Score of ≥ 4 for at least 2 of the following PANSS items: delusions (P1), conceptual disorganization (P2), hallucinatory behavior (P3), suspiciousness (P6), somatic concern (G1), or unusual thought content (G9) at screening visit
* Score ≥ 4 (at least moderately ill) on the Clinical Global Impression of Severity (CGI-S) at screening visit.
* Undergoing treatment with at least 1 antipsychotic medication with no change in dosing, supported by documentation, for at least 8 weeks prior to screening and no change in antipsychotic medication dosing planned throughout the trial
* Taking a maximum of 2 antipsychotic medications. For participants taking oral antipsychotic medications only, the sum of primary and secondary antipsychotic medications is ≤ 30 milligrams (mg)/day of oral olanzapine equivalents. For participants taking long-acting injectable antipsychotic medications, the dose is within the range approved and any secondary oral antipsychotic medications is ≤ 5 mg/day of oral olanzapine equivalents.
* Documented response (at least partially) to treatment with current antipsychotic medications (e.g., treatment of recent exacerbation of psychotic symptoms)
* On a stable dose if taking concomitant psychotropic medications and within allowed limits, including antidepressants, anxiolytics, anticholinergics and/or antiepileptics for at least 4 weeks prior to screening (dose reductions ≤ 25% of total dose are permitted) with no plans to change dosing during the trial (i.e., from screening onwards). Valproic acid or any prescribed valproate product (valproate semisodium or valproate sodium) is disallowed within 4 weeks (i.e., more than 5 half lives) prior to the baseline visit.

Exclusion Criteria:

Diagnosis and Psychiatric History

* Recent (within the last 3 months prior to screening) diagnosis of panic disorder, depressive episode, or other comorbid psychiatric conditions based on the MINI for Psychotic Disorders Studies (or DSM-5) OR has PANSS item G6 score of ≥ 5 (depression) at screening.
* Any psychiatric disorder that may interfere with the conduct of this trial, including but not limited to attention deficit hyperactivity disorder, pervasive developmental disorder, intellectual disability, personality disorder that might interfere with compliance or increase suicidal risk, manic or hypomanic episode, or any other psychotic disorder, as defined in the DSM-5
* Current diagnosis or a history of substance use disorder according to DSM-5 criteria within 6 months prior to screening or prior chronic substance abuse judged likely to recur during the trial period by the investigator. Nicotine use or occasional cannabis use (≤ 3 days per week recreational cannabis use) is acceptable. Corroboration of the participant's frequency of cannabis use by an adult informant (e.g., family member, social worker, caseworker, residential facility staff, or nurse), should be obtained if the participant has a positive urine test for Δ9-tetrahydrocannabinol at screening.
* A positive drug screen for opiates, methadone, cocaine, amphetamines (including ecstasy), or barbiturates; a repeat drug screen may be done to verify the result.
* Any history of suicidal behavior or any suicidal ideation of type 4 or 5 on the adult C-SSRS or within 1 month prior to screening

Treatment History

* Treatment-resistant schizophrenia as judged by the treating physician and as defined by having previously demonstrated no response to > 2 trials of antipsychotic trial medications at therapeutic doses or required clozapine therapy due to non-response to antipsychotic therapy within the previous 6 months.
* Based on the investigator assessment, current antipsychotic medication blood levels are below the therapeutic range if therapeutic drug monitoring is available for the antipsychotic(s) prescribed for the participant; or there is no documentation confirming the administration of long-acting injectable antipsychotic medication within the approved dose range and as prescribed by the treating physician.

Past and Current Medical History

* History of moderate or severe head trauma (for example, loss of consciousness for more than 15 minutes) or other neurological disorders (including epilepsy), neurodegenerative disorder (Alzheimer's disease, Parkinson's disease, multiple sclerosis, Huntington's disease, etc.) or systemic medical diseases that are, in the opinion of the investigator, likely to interfere with the conduct of the trial or confound the trial assessments
* Tardive dyskinesia (TD) that is moderate to severe (i.e., a score of > 21 on the dyskinesia subscale of the Extrapyramidal Symptom Rating Scale [ESRS] at screening) or requires treatment
* Any other significant disease, disorder, pending court proceedings or social circumstances which, in the opinion of the investigator, may either put the participant at risk because of participation in the trial, may influence the result of the trial, or may affect the participant's ability to take part in the trial.

Other

* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the investigational medicinal product, such as sesame seed oil
* One or more laboratory values outside the normal range, based on the blood or urine samples taken at the screening visit, that are considered by the investigator to be clinically significant; or impaired hepatic function at screening, defined as serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN) or total bilirubin (TBL) > 1.5 × ULN or international normalized ratio (INR) > 1.2 (TBL ULN parameter not applicable for participants diagnosed with Gilbert's disease)
* Currently using or within 3 months of screening has used cannabidiol (CBD) oil or purified CBD preparations and is unwilling to abstain for the duration of the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (19):
  - Clinical Trial Site, Bentonville, Arkansas
  - Clinical Trial Site, Little Rock, Arkansas
  - Clinical Trial Site, Garden Grove, California
  - Clinical Trial Site, Lemon Grove, California
  - Clinical Trial Site, Oakland, California
  - Clinical Trial Site, Pico Rivera, California
  - Clinical Trial Site, Largo, Florida
  - Clinical Trial Site, Lauderhill, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Lincolnwood, Illinois
  - Clinical Trial Site, Shreveport, Louisiana
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, Berlin, New Jersey
  - Clinical Trial Site, Cedarhurst, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Rochester, New York
  - Clinical Trial Site, Beachwood, Ohio
  - Clinical Trial Site, Richardson, Texas
- Poland (7):
  - Clinical Trial Site, Bełchatów
  - Clinical Trial Site, Gdansk
  - Clinical Trial Site, Kielce
  - Clinical Trial Site, Kobierzyce
  - Clinical Trial Site, Poznan
  - Clinical Trial Site, Torun
  - Clinical Trial Site, Wroclaw
- Serbia (8):
  - Clinical Trial Site#1, Belgrade
  - Clinical Trial Site#2, Belgrade
  - Clinical Trial Site#1, Kovin
  - Clinical Trial Site#2, Kovin
  - Clinical Trial Site#1, Kragujevac
  - Clinical Trial Site#2, Kragujevac
  - Clinical Trial Site#3, Kragujevac
  - Clinical Trial Site, Niš
- Spain (4):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Oviedo
  - Clinical Trial Site, Salamanca
  - Clinical Trial Site, Valladolid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 95 participants who met all inclusion and no exclusion criteria were enrolled in the study and were randomized to the Placebo Run-in Period. Eighteen participants failed the Placebo Run-in Period. A total of 77 participants were randomized to 1 of 2 GWP42003-P doses or placebo treatment at a 2:2:1:1 ratio at 33 clinic centers.
Pre-assignment Details: Once enrolled, participants were randomized to treatment following a single-blind, 2-week Placebo Run-in Period. A total of 95 participants were included the Placebo Run-in Period; 18 participants failed the Placebo Run-in Period. A total of 77 participants were randomized to the Treatment Period.
Groups:
- GWP42003-P 300 mg: Clinically stable schizophrenia participants experiencing inadequate response to antipsychotic treatment who were randomized to receive an oral dose of GWP42003-P 300 milligrams (mg) per day for 12 weeks.
- GWP42003-P 1000 mg: Clinically stable schizophrenia participants experiencing inadequate response to antipsychotic treatment who were randomized to receive an oral dose of GWP42003-P 1000 milligrams (mg) per day for 12 weeks.
- Pooled Placebo: Clinically stable schizophrenia participants experiencing inadequate response to antipsychotic treatment who were randomized to receive a matching placebo per day for 12 weeks.
Period: Randomized Placebo Run-in Period
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Started | 0 | 0 | 95
Completed | 0 | 0 | 77
Not Completed | 0 | 0 | 18
Not completed — Placebo Run-in Failures | 0 | 0 | 18
Period: Randomized Treatment Period
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Started | 27 (Of the 77 participants who completed the Placebo Run-in Period, 27 were randomized to GWP42003-P 300 mg.) | 24 (Of the 77 participants who completed the Placebo Run-in Period, 24 were randomized to GWP42003-P 1000 mg.) | 26 (Of the 77 participants who completed the Placebo Run-in Period, 26 were randomized to pooled placebo.)
Completed | 23 | 19 | 19
Not Completed | 4 | 5 | 7
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal of parent/legal representative consent | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Participant non-compliance | 1 | 1 | 2
Not completed — Other | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics were assessed in the Full Analysis Set in the Treatment Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo | Total
Number analyzed (Participants) | 27 | 24 | 26 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 24 | 26 | 77
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (7.53) | 39.2 (8.21) | 38.7 (8.87) | 38.4 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 7 | 20
  Male | 21 | 17 | 19 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 11 | 7 | 10 | 28
  White | 15 | 17 | 14 | 46
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 14 | 18 | 52
  Poland | 1 | 1 | 1 | 3
  Serbia | 6 | 8 | 6 | 20
  Spain | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Least Square Mean Change From Baseline in the Positive and Negative Symptoms Scale (PANSS) Total (PANSS-T) Score
Description: The PANSS-T is a medical scale used for measuring symptom severity of participants with schizophrenia or related psychotic disorder. It is a 30-item rating instrument that assesses the positive and negative symptoms of schizophrenia as well as symptoms of general psychopathology. Individual items are rated on a 7-point scale, where 1 = absent and 7 = extreme. A PANSS-T score is derived from the sum of the 30 items and the total score ranges from 30 to 210, where higher scores represent worse outcome. The least square mean change from baseline is being reported and negative values indicate an improvement in outcome.
Time Frame: Baseline up to Week 12
Population: Efficacy outcomes were assessed in the Full Analysis Set in participants with available data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
units on a scale | -10.49 (1.64) | -10.69 (1.75) | -8.74 (1.78)
Statistical Analysis 1: Comparison: GWP42003-P 300 mg vs Pooled Placebo; Test type: Superiority — The repeated measures model includes stratification factors (sex and region), associated baseline, visit, randomised treatment arm and visit by treatment arm interaction as fixed effects and visit repeated within each participant as a repeated effect. For the PANSS-T score, baseline PANSS-P, baseline PANSS-N, and baseline PANSS-G are included in the model as fixed effects for the associated baseline instead of baseline PANSS-T; p = 0.4528, Mixed-effects repeated measures model; Least square mean difference = -1.75, 95% CI 2-sided [-6.35 to 2.84], Standard Error of Mean 2.33
Statistical Analysis 2: Comparison: GWP42003-P 1000 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4226, Mixed-effects repeated measures model; Least square mean difference = -1.96, 95% CI 2-sided [-6.76 to 2.85], Standard Error of Mean 2.44

2. Primary Outcome: Least Square Mean Change From Baseline in the PANSS Positive Subscale (PANSS-P) Score
Description: The PANSS 'P' Scale was calculated as the sum of the items prefixed with an P, 7 items in total, i.e. delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution and hostility. Individual items are rated on a 7-point scale, where 1 = absent and 7 = extreme. The least square mean change from baseline is being reported and negative values indicate an improvement in outcome.
Time Frame: Baseline up to Week 12
Population: Efficacy outcomes were assessed in the Full Analysis Set in participants with available data.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
units on a scale | -3.16 (0.59) | -3.75 (0.63) | -2.53 (0.62)
Statistical Analysis 1: Comparison: GWP42003-P 300 mg vs Pooled Placebo; Test type: Superiority — The repeated measures model includes stratification factors (sex and region), associated baseline, visit, randomised treatment arm and visit by treatment arm interaction as fixed effects and visit repeated within each participant as a repeated effect; p = 0.4479, Mixed-effects repeated measures model; Least square mean difference = -0.63, 95% CI 2-sided [-2.25 to 1.00], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: GWP42003-P 1000 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.1616, Mixed-effects repeated measures model; Least square mean difference = -1.22, 95% CI 2-sided [-2.92 to 0.49], Standard Error of Mean 0.87

3. Primary Outcome: Least Square Mean Change From Baseline in the PANSS Negative Subscale (PANSS-N) Score
Description: The PANSS 'N' Scale will be calculated as the sum of the items prefixed with an N, 7 items in total, i.e. blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation and stereotyped thinking. Individual items are rated on a 7-point scale, where 1 = absent and 7 = extreme. The least square mean change from baseline is being reported and negative values indicate an improvement in outcome.
Time Frame: Baseline up to Week 12
Population: Efficacy outcomes were assessed in the Full Analysis Set in participants with available data.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
units on a scale | -2.64 (0.53) | -1.57 (0.56) | -2.33 (0.58)
Statistical Analysis 1: Comparison: GWP42003-P 300 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6787, Mixed-effects repeated measures model; Least square mean difference = -0.31, 95% CI 2-sided [-1.80 to 1.18], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: GWP42003-P 1000 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.3351, Mixed-effects repeated measures model; Least square mean difference = 0.76, 95% CI 2-sided [-0.79 to 2.30], Standard Error of Mean 0.78

4. Primary Outcome: Least Square Mean Change From Baseline in the PANSS General Subscale (PANSS-G) Score
Description: The PANSS 'G' Scale will be calculated as the sum of the items prefixed with a G, 16 items in total, i.e. somatic concerns, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation and active social avoidance. Individual items are rated on a 7-point scale, where 1 = absent and 7 = extreme. The least square mean change from baseline is being reported and negative values indicate an improvement in outcome.
Time Frame: Baseline up to Week 12
Population: Efficacy outcomes were assessed in the Full Analysis Set in participants with available data.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
units on a scale | -4.78 (1.03) | -4.91 (1.10) | -3.68 (1.09)
Statistical Analysis 1: Comparison: GWP42003-P 300 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.4504, Mixed-effects repeated measures model; Least square mean difference = -1.10, 95% CI 2-sided [-3.96 to 1.76], Standard Error of Mean 1.45
Statistical Analysis 2: Comparison: GWP42003-P 1000 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.4195, Mixed-effects repeated measures model; Least square mean difference = -1.23, 95% CI 2-sided [-4.22 to 1.76], Standard Error of Mean 1.52

5. Primary Outcome: Least Square Mean Change From Baseline in the Clinical Global Impression of Severity (CGI-S) Score
Description: The CGI-S is a 7-point scale used to rate the severity of participants' illness at the time of assessment. Considering total clinical experience, a participant will be assessed on severity of mental illness at the time of rating 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = among the most extremely ill participants. The least square mean change from baseline is being reported and negative values indicate an improvement in outcome.
Time Frame: Baseline up to Week 12
Population: Efficacy outcomes were assessed in the Full Analysis Set.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
units on a scale | -0.47 (0.11) | -0.50 (0.12) | -0.45 (0.12)
Statistical Analysis 1: Comparison: GWP42003-P 300 mg vs Pooled Placebo; Test type: Superiority — The repeated measures model includes stratification factors (sex and region), associated baseline, visit, randomised treatment arm, visit by treatment arm interaction and visit by associated baseline interaction as fixed effects and visit repeated within each participant as a repeated effect; p = 0.8850, Mixed-effects repeated measures model; Least square mean difference = 0.02, 95% CI 2-sided [-0.35 to 0.30], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: GWP42003-P 1000 mg vs Pooled Placebo; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.7808, Mixed-effects repeated measures model; Least square mean difference = 0.04, 95% CI 2-sided [-0.36 to 0.27], Standard Error of Mean 0.16

6. Primary Outcome: Number of Participants With Minimally or Better Clinical Global Impression of Improvement (CGI-I) Score at Week 12
Description: The CGI-I is a 7-point scale used to rate the improvement of participants' condition at the time of assessment. Compared to the patient's condition at baseline, the participants' condition was rated as 1 = very much improved since initiation of treatment; 2 = much improved; 3 = minimally improved; 4 = no change from baseline; 5 = minimally worse; 6 = much worse; 7 = very much worse since the initiation of treatment. Higher scores indicate a worse outcome. The number of participants with minimally or better improvements (score of 3 or better) are being reported.
Time Frame: Week 12
Population: Clinical Global Impression of Improvement (CGI-I) Score was assessed in the Full Analysis Set in participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
Participants | 17 | 12 | 15
Statistical Analysis 1: Comparison: GWP42003-P 300 mg vs Pooled Placebo; Test type: Superiority; p = 0.6707, Regression, Logistic; Odds Ratio (OR) = 1.412, 95% CI 2-sided [0.288 to 6.924]
Statistical Analysis 2: Comparison: GWP42003-P 1000 mg vs Pooled Placebo; Test type: Superiority; p = 0.4883, Regression, Logistic; Odds Ratio (OR) = 0.576, 95% CI 2-sided [0.121 to 2.744]

7. Secondary Outcome: Mean Change From Baseline in Body Weight
Time Frame: Baseline up to Week 12
Population: Body weight was assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
kilogram | -0.03 (3.09) | -0.14 (1.98) | 1.37 (1.28)

8. Secondary Outcome: Mean Change From Baseline in Body Mass Index (BMI)
Time Frame: Baseline up to Week 12
Population: Body mass index was assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
kg/m^2 | 0 (0.98) | -0.04 (0.66) | 0.45 (0.45)

9. Secondary Outcome: Mean Change From Baseline in Waist Circumference
Time Frame: Baseline up to Week 12
Population: Waist circumference was assessed in the Safety Analysis set in participants with available data.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
centimeters | 0.41 (5.36) | -0.53 (2.07) | 1.34 (3.13)

10. Secondary Outcome: Mean Change From Baseline in Blood Pressure
Time Frame: Baseline up to Week 12
Population: Blood pressure was assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
mmHg
  Diastolic blood pressure | 1.7 (6.19) | 0 (7.05) | -0.2 (5.71)
  Systolic blood pressure | 0.3 (9.38) | 0 (8.41) | 0.3 (5.66)

11. Secondary Outcome: Mean Change From Baseline in Heart Rate
Time Frame: Baseline up to Week 12
Population: Heart rate was assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
beats/minute | 1.0 (8.46) | -3.1 (9.13) | 0.1 (6.52)

12. Secondary Outcome: Mean Change From Baseline in Respiratory Rate
Time Frame: Baseline up to Week 12
Population: Respiratory rate was assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
breaths/minute | -0.6 (2.13) | 0.1 (1.37) | 0 (1.45)

13. Secondary Outcome: Mean Change From Baseline in Temperature
Time Frame: Baseline up to Week 12
Population: Temperature was assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
Celsius | -0.07 (0.34) | 0.06 (0.20) | -0.02 (0.19)

14. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Test Results
Time Frame: Day 85
Population: Clinically significant changes from baseline in vital signs were assessed in the Safety Analysis Set in participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 23 | 19 | 19
Participants
  Supine systolic blood pressure, Day 85: <-20 | 0 | 0 | 0
  Supine systolic blood pressure, Day 85: >20 | 1 | 0 | 0
  Supine diastolic blood pressure, Day 85: <-10 | 0 | 1 | 0
  Supine diastolic blood pressure, Day 85: >10 | 2 | 1 | 0
  Heart rate, Day 85: <-20 | 0 | 0 | 0
  Heart rate, Day 85: >20 | 0 | 0 | 0
  Weight, Day 85: ≤-7% | 2 | 1 | 0
  Weight, Day 85: ≥7% | 1 | 0 | 0

15. Secondary Outcome: Number of Participants With Defined Flagged Electrocardiogram (ECG) Parameter Values
Time Frame: Day 85
Population: Defined flagged ECG values were assessed in the Safety Analysis Set in participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 27 | 24 | 26
Participants
  QTcF interval, Day 85: >450 msec | 0 | 1 | 0
  QTcF interval, Day 85: >480 msec | 0 | 0 | 0
  QTcF interval, Day 85: >500 msec | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior Based on The Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a short questionnaire that is used to assess suicidal ideation (5 questions) and behavior (5 questions) since last patient visit. The questionnaire is completed by participants answering yes or no to each question.
Time Frame: Baseline (screening) up to Day 85
Population: Suicidal ideation and behavior was assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo
Number analyzed (Participants) | 24 | 27 | 26
Participants
  Screening, Suicidal ideation, Wish to be dead | 1 | 0 | 0
  Screening, Suicidal ideation, Non-specific active suicidal thoughts | 0 | 0 | 0
  Screening, Suicidal ideation, Active with any methods (not planned) without intent to act | 0 | 0 | 0
  Screening, Suicidal ideation, Active with some intent to act, without specific plan | 0 | 0 | 0
  Screening, Suicidal ideation, Active with specific plan and intent | 0 | 0 | 0
  Screening, Suicidal behavior, Preparatory acts or behavior | 0 | 0 | 0
  Screening, Suicidal behavior, Aborted attempt | 0 | 0 | 0
  Screening, Suicidal behavior, Interrupted attempt | 0 | 0 | 0
  Screening, Suicidal behavior, Actual attempt | 0 | 0 | 0
  Screening, Suicidal behavior, Completed suicide | 0 | 0 | 0
  Day 14, Suicidal ideation, Wish to be dead | 0 | 1 | 0
  Day 14, Suicidal ideation, Non-specific active suicidal thoughts | 0 | 0 | 0
  Day 14, Suicidal ideation, Active with any methods (not planned) without intent to act | 0 | 0 | 0
  Day 14, Suicidal ideation, Active with some intent to act, without specific plan | 0 | 0 | 0
  Day 14, Suicidal ideation, Active with specific plan and intent | 0 | 0 | 0
  Day 14, Suicidal behavior, Preparatory acts or behavior | 0 | 0 | 0
  Day 14, Suicidal behavior, Aborted attempt | 0 | 0 | 0
  Day 14, Suicidal behavior, Interrupted attempt | 0 | 0 | 0
  Day 14, Suicidal behavior, Actual attempt | 0 | 0 | 0
  Day 14, Suicidal behavior, Completed suicide | 0 | 0 | 0
  Day 29, Suicidal ideation, Wish to be dead | 1 | 1 | 0
  Day 29, Suicidal ideation, Non-specific active suicidal thoughts | 0 | 1 | 0
  Day 29, Suicidal ideation, Active with any methods (not planned) without intent to act | 0 | 1 | 0
  Day 29, Suicidal ideation, Active with some intent to act, without specific plan | 0 | 0 | 0
  Day 29, Suicidal ideation, Active with specific plan and intent | 0 | 0 | 0
  Day 29, Suicidal behavior, Preparatory acts or behavior | 0 | 0 | 0
  Day 29, Suicidal behavior, Aborted attempt | 0 | 0 | 0
  Day 29, Suicidal behavior, Interrupted attempt | 0 | 0 | 0
  Day 29, Suicidal behavior, Actual attempt | 0 | 0 | 0
  Day 29, Suicidal behavior, Completed suicide | 0 | 0 | 0
  Day 85, Suicidal ideation, Wish to be dead | 0 | 0 | 0
  Day 85, Suicidal ideation, Non-specific active suicidal thoughts | 0 | 0 | 0
  Day 85, Suicidal ideation, Active with any methods (not planned) without intent to act | 0 | 0 | 0
  Day 85, Suicidal ideation, Active with some intent to act, without specific plan | 0 | 0 | 0
  Day 85, Suicidal ideation, Active with specific plan and intent | 0 | 0 | 0
  Day 85, Suicidal behavior, Preparatory acts or behavior | 0 | 0 | 0
  Day 85, Suicidal behavior, Aborted attempt | 0 | 0 | 0
  Day 85, Suicidal behavior, Interrupted attempt | 0 | 0 | 0
  Day 85, Suicidal behavior, Actual attempt | 0 | 0 | 0
  Day 85, Suicidal behavior, Completed suicide | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from baseline up to end of study, approximately 1 year 8 months.
Groups:
- Pooled Placebo (Treatment Period): Clinically stable schizophrenia participants experiencing inadequate response to antipsychotic treatment who were randomized to receive a matching placebo per day for 12 weeks.
- Pooled Placebo (Placebo Run-In Period): Clinically stable schizophrenia participants experiencing inadequate response to antipsychotic treatment who were randomized to receive a matching placebo for 2 weeks (including participants who failed the placebo-run in period).
Arm/Group | GWP42003-P 300 mg | GWP42003-P 1000 mg | Pooled Placebo (Treatment Period) | Pooled Placebo (Placebo Run-In Period)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/24 | 0/26 | 0/95
Serious Adverse Events (participants affected / at risk) | 2/27 | 2/24 | 1/26 | 0/95
Other Adverse Events (participants affected / at risk) | 3/27 | 3/24 | 3/26 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 300 mg (N=27) | GWP42003-P 1000 mg (N=24) | Pooled Placebo (Treatment Period) (N=26) | Pooled Placebo (Placebo Run-In Period) (N=95)
COVID-19 (Infections and infestations) | 2 | 0 | 0 | NA
Coronavirus infection (Infections and infestations) | 0 | 1 | 0 | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA
Hospitalization (Surgical and medical procedures) | 0 | 0 | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 300 mg (N=27) | GWP42003-P 1000 mg (N=24) | Pooled Placebo (Treatment Period) (N=26) | Pooled Placebo (Placebo Run-In Period) (N=95)
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT04421456/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT04421456/SAP_001.pdf